CLINICAL TRIAL: NCT07163351
Title: Prefabricated CAD CAM Allogeneic Ring Blocks in the Anterior Maxilla With Immediate Implantation a Prospective Single-Arm Clinical Study
Brief Title: Prefabricated CAD CAM Allogeneic Ring Blocks in the Anterior Maxilla With Immediate Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Omar Elboraey Elbal, Assistant Professor of Oral Medicine, Periodontology, Oral Diagnosis and Oral Radiology Department, Faculty of Dentistry, Tanta, University, Tanta, Egypt., Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUAREC20240001-7
Record Dates: First submitted 2025-08-31; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Prefabricated; CAD; CAM; Allogeneic Ring Blocks; Anterior Maxilla; Immediate Implantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Patients presented with anterior maxillary alveolar bone defects resulting from previous implant failure
  Interventions: Other: CAD/CAM allogenic bone block

INTERVENTIONS:
Other: CAD/CAM allogenic bone block — CAD/CAM allogenic bone block augmentation with immediate non-functional implant loading

SUMMARY:
Clinical and radiographic evaluation of a new modification of ring technique using omputeraided design/computer-aided manufacturing (CAD/CAM) milling of allogeneic bone block for anterior maxilla ridge augmentation with immediate implantation

DETAILED DESCRIPTION:
Dental implant failure remains a clinically significant challenge, with early failures typically attributed to insufficient osseointegration, surgical trauma, bacterial contamination, or micromotion during healing. In contrast, late failures are often associated with occlusal overload, peri-implantitis, or implant mispositioning.

These challenges have driven the adoption of allogeneic bone blocks, particularly those fabricated using computeraided design/computer-aided manufacturing (CAD/CAM) technology, which offer precise anatomical adaptation, reduced surgical time, and minimized complications compared to manual grafting techniques

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years.
* Both sexes.
* Patients presenting with anterior maxillary alveolar bone defects resulting from previous implant failure.
* Systemically healthy individuals, classified as American Society of Anesthesiologists (ASA) physical status I or II.
* Participants were either non-smokers or light smokers consuming fewer than 10 cigarettes per day.

Exclusion Criteria:

* Uncontrolled systemic conditions such as diabetes mellitus or osteoporosis.
* Pregnant or breastfeeding at the time of recruitment.
* Individuals with a history of head or neck radiation therapy.
* Cases in which insufficient bone volume for implant placement persisted following augmentation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Vertical/Horizonal Bone Gain | 18 months post-procedure
  Vertical/Horizonal Bone Gain was measured via cone beam computed tomography superimposition at 18 months

SECONDARY OUTCOMES:
Implant Survival Rate | 18 months post-procedure
  Implant survival rate, defined as the absence of clinical mobility, peri-implant infection, persistent pain, or radiographic evidence of peri-implant radiolucency or bone loss beyond expected physiological remodelling. Implant stability was assessed clinically using percussion and mobility tests, and radiographically using periapical radiographs and/or cone-beam computed tomography at designated follow-up intervals. Survival was evaluated at 6, 12, and 18 months postoperatively
Assessment of aesthetic outcome | 18 months post-procedure
  Assessment of aesthetic outcome were assessed using the Pink Esthetic Score (PES), a validated clinical index that evaluates seven soft tissue parameters around the implant site: mesial and distal papillae, soft tissue level, soft tissue contour, alveolar process deficiency, soft tissue color, and texture. PES was evaluated at 12 and 18 months by two calibrated examiners blinded to the treatment allocation.
Patient Satisfaction | 18 months post-procedure
  Patient-reported satisfaction with the aesthetic and functional outcomes was measured using a 10-point Visual Analog Scale (VAS). Patients were asked to rate their satisfaction with the final restoration, including perceived appearance, comfort, and chewing efficiency at 12 and 18 months postoperatively. Mean VAS scores were analyzed and compared over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.